CLINICAL TRIAL: NCT03606889
Title: Quadratus Lumborum Block vs Transversus Abdominis Plane Block for Post-prostatectomy Analgesia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not enough participants
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Tomasz Skladzien, MD PHD, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1072.6120.107.2018
Record Dates: First submitted 2018-07-11; First posted 2018-07-31 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Prostatic Cancer; Pain, Postoperative; Pain; Anesthetics, Local
MeSH Terms: conditions — Prostatic Neoplasms; Pain, Postoperative; Pain | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quadratus Lumborum block group (Experimental): Quadratus Lumborum block group (QL) patients will receive a bilateral Quadratus Lumborum block using Bupivicaine 0.125%
  Interventions: Diagnostic Test: Quadratus Lumborum block; Drug: Bupivacaine
- Transversus abdominis plane block group (Experimental): Transversus abdominis plane block (TAP) patients will receive a bilateral TAP block using Bupivicaine 0.125%
  Interventions: Diagnostic Test: Tranversus Abdominis plane block; Drug: Bupivacaine

INTERVENTIONS:
Diagnostic Test: Quadratus Lumborum block — 0.2 ml/kg bupivicaine 0.125% injected bilateraly at the posterior border of the quadratus Lumborum muscle
  Other Names: QLB
  Arms: Quadratus Lumborum block group
Diagnostic Test: Tranversus Abdominis plane block — 0.2 ml/kg bupivicaine 0.125% injected bilateraly between internal oblique and transversus abdominis muscles.
  Other Names: TAP
  Arms: Transversus abdominis plane block group
Drug: Bupivacaine — 0.2 ml/kg bupivicaine

SUMMARY:
Recently, the uses of peripheral axial blocks that deliver local anesthetic into the transversus abdominis fascial plane have become popular for operations that involve incision(s) of the abdominal wall. Thus, the Transversus Abdominis plane (TAP) block has been shown to reduce perioperative opioid use in elective abdominal surgery, including open appendicectomy, laparotomy, and laparoscopic cholecystectomy.

Currently, the Quadratus Lumborum block (QL block) is performed as one of the perioperative pain management procedures for all generations (pediatrics, pregnant, and adult) undergoing abdominal surgery. The local anesthetic injected via the approach of the posterior QL block ( QL 2 block ) can more easily extend beyond the TAP to the thoracic paravertebral space or the thoracolumbar plane, the posterior QL block entails a broader sensory-level analgesic and may generate analgesia from T7 to L1. Use of posterior QL block in laparoscopic prostatectomy has not been investigated before and it is the variant that will be discussed in our study.

DETAILED DESCRIPTION:
In laparoscopic prostatectomy, overall pain is a conglomerate of three different and clinically separate components: incisional pain (somatic pain), visceral pain (deep intra abdominal pain), and shoulder pain due to peritoneal stretching and diaphragmatic irritation associated with carbon dioxide insufflation. Moreover, it has been hypothesized that intense acute pain after laparoscopic prostatectomy may predict development of chronic pain. Without effective treatment, this ongoing pain may delay recovery, mandate inpatient admission, and thereby increase the cost of such care.

ELIGIBILITY:
Inclusion Criteria:

* Pateints who will have prostatectomy ASA II or III

Exclusion Criteria: Patient refusal Local infection at the site of injection Allergy to study medications Sepsis Anatomic abnormalities Systemic anticoagulation or coagulopathy Inability to comprehend or participate in pain scoring system Inability to use intravenous patient controlled analgesia

-

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate is only in males.
Enrollment: 12 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Total oxycodone used in the first 24 hours after surgery | 24 hours
  Total cumulative oxycodone dose in mg used in the first 24 hours after surgery

SECONDARY OUTCOMES:
Severity of postoperative pain via visual analogue pain scale (VAS) | 24 hours
  VAS range from 0 for no pain to 10 for worst pain imaginable

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Skladzien, MD PHD, Principal Investigator — Jagiellonian University
Locations (1):
- University Hospital in Cracow, Krakow, Poland

IPD SHARING:
Plan to Share IPD: Undecided